CLINICAL TRIAL: NCT04421911
Title: A Study to Comparing the Efficacy and Safety of the Ketoprofen and Diclofenac in Patients With Osteoarthritis
Brief Title: A Study to Assess Efficacy and Safety of the Ketoprofen vs Diclofenac
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KETO-2019
Record Dates: First submitted 2020-06-02; First posted 2020-06-09 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Osteoarthritis
Keywords: ketoprofen; diclofenac; osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Ketoprofen; Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketoprofen (Experimental)
  Interventions: Drug: Ketoprofen topical
- Diclofenac (Active Comparator)
  Interventions: Drug: Diclofenac Topical

INTERVENTIONS:
Drug: Ketoprofen topical — Ketoprofen topical for 21days
  Arms: ketoprofen
Drug: Diclofenac Topical — Diclofenac topical for 21days
  Arms: Diclofenac

SUMMARY:
Primary objective:

• To assess therapeutic efficacy of the Ketoprofen compared with Diclofenac based on the assessment of primary endpoint : Mean change in walking arthritis pain intensity score

Secondary objectives:

* To assess therapeutic efficacy of the Ketoprofen compared with Diclofenac based on the assessment of secondary endpoints.
* To assess safety and tolerability of the Ketoprofen compared with Diclofenac based on the nature and frequency of adverse events in treatment groups

DETAILED DESCRIPTION:
This trial is designed as an open-label, multicenter, randomized, clinical study for assessment of efficacy and safety of Ketoprofen plaster and Diclofenac plaster in patients with osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40-75 years
* Compliance to ACR diagnostic criteria of OA of the knee
* Patients with Kellgren-Lawrence grade 1-3
* Index knee pain should be ≥40 mm on VAS (100mm) scale

Exclusion Criteria:

* Intolerance or allergic reactions to the study therapy
* Usage of NSAIDs within 3 days
* Open skin lesions or dermatological conditions at the site of plaster application
* Surgery or major trauma of the index knee within the previous 12 months
* Pregnant or breast-feeding women
* Alcohol addiction, drug addiction or drug abuse in the past

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Mean change in walking arthritis pain intensity score | 3 weeks
  Pain will be assessed by a horizontal 100 mm Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Mean change in spontaneous arthritis pain intensity score | 3 weeks
  Pain will be assessed by a horizontal 100 mm Visual Analogue Scale (VAS)
Knee injury and Osteoarthritis Outcome Score (KOOS) | 3 weeks
  Mean change in individual parameters and the general normalized Knee injury and Osteoarthritis Outcome Score (KOOS) score (5-point scale)
Global Impression of Improvement (PGI-I) | 3 weeks
  Patient Global Impression of Improvement (PGI-I) assessment
Adverse events | 3 weeks
  frequency, severity, relationship with the study drug

CONTACTS AND LOCATIONS:
Locations (9):
- Russia (9):
  - Maksimum Zdorovya, Kemerovo
  - City Clinical Hospital #1 n.a. Pirogova, Moscow
  - Rostov State Medical University, Rostov-on-Don
  - Ryazan State Medical University n.a. I.P.Pavlov, Ryazan
  - Saratov State Medical University n.a. V.I.Razumovsky, Saratov
  - Private Healthcare Institution Smolensk Russian Railway Clinical Hospital, Smolensk
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk
  - Regional Clinical Hospital, Vladimir
  - Clinical Emergency Hospital n.a. N.V.Soloviev, Yaroslavl

IPD SHARING:
Plan to Share IPD: No